CLINICAL TRIAL: NCT07095582
Title: Enhancing Therapist-Guided Internet-Delivered Cognitive Behaviour Therapy for Depression and Anxiety With Additional Content
Brief Title: Enhancing Internet-Delivered Cognitive Behaviour Therapy With Additional Content
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: Government of Saskatchewan, Ministry of Health (Unknown); Linkoeping University (Other Government); Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1086
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Loneliness; Depression; Anxiety
Keywords: Loneliness; Depression; Anxiety; Internet-delivered cognitive behavioral therapy; Randomized controlled trial; Personalized therapy; Therapist assistance; Mental health system
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellbeing Course (No Loneliness Content) (Active Comparator): All clients eligible for ICBT will be screened for frequent loneliness. Due to practical constraints related to therapist workload and the volume of referrals, a subset of eligible clients scoring ≥ 6 on the UCLA loneliness scale, will be randomly assigned to the Wellbeing Course or the Wellbeing Course plus Loneliness Content. Participants in both conditions will receive the Wellbeing Course which consists of 5 ICBT lessons released gradually over 8 weeks. They will also receive 8 weeks of therapist support, with the option of extending support to 12 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy
- Wellbeing Course plus Loneliness Content (Experimental): Due to practical constraints related to therapist workload and the volume of referrals, a subset of eligible clients scoring ≥ 6 on the UCLA loneliness scale, will be randomly assigned to the Wellbeing Course or the Wellbeing Course plus Loneliness Content. In the Loneliness Content condition, in addition to the 5 ICBT lessons from the Wellbeing Course, participants will receive content pertaining to loneliness with each lesson. This content will be presented at the end of each new lesson of the Wellbeing Course, and provide psychoeducation on loneliness and skills for addressing loneliness. Participants in the Loneliness Content condition will also receive 8 weeks of therapist support, with the option of extending support to 12 weeks.
  Interventions: Behavioral: Internet-delivered cognitive behavioral therapy; Behavioral: Additional Loneliness Content

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioral therapy — The Wellbeing Course was developed at Macquarie University, Australia. The Wellbeing Course is a transdiagnostic Internet-delivered cognitive behavioural intervention targeting symptoms of depressive and anxiety disorders. It comprises 5 online lessons targeting: 1) symptom identification and the cognitive behavioural model; 2) thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling; 4) graduated exposure; and 5) relapse prevention. Materials are presented in a didactic (i.e., text-based with visual images) and case-enhanced learning format (i.e., educational stories demonstrate the application of skills) and include homework activities. Lessons are released gradually in a standardized order over 8 weeks. Phone calls will only be made if there is a significant clinical issue requiring therapist attention that cannot be addressed over email (e.g., sudden increase in symptoms). Therapists will spend ~15 mins per week/per client.
Behavioral: Additional Loneliness Content — The additional Loneliness Content was developed at the Online Therapy Unit, University of Regina, Canada. Relevant sections of the resource will be included at the end of each lesson within the Wellbeing Course. The Loneliness Content provides psychoeducation and skills for loneliness using a cognitive behavioral framework. Consistent with the Wellbeing Course content, the Loneliness Content will target 1) identification of loneliness; 2) loneliness thought monitoring and challenging; 3) de-arousal strategies and pleasant activity scheduling for loneliness; 4) behaviours (conversation skills); and 5) relapse prevention.
  Arms: Wellbeing Course plus Loneliness Content

SUMMARY:
This study evaluates the effectiveness of additional content on loneliness offered alongside the Wellbeing Course - an internet-delivered cognitive behavioral therapy (ICBT) intervention for symptoms of depression and anxiety- in improving treatment outcomes for individuals with elevated scores on loneliness seeking treatment for depression and anxiety at a routine care online therapy clinic (the Online Therapy Unit). In this partially randomized control trial, the investigators aim to contribute to the literature by examining whether providing additional content on loneliness alongside the Wellbeing Course enhances engagement, satisfaction, and treatment outcomes among clients experiencing frequent loneliness compared to those completing only the Wellbeing Course. Over 8 weeks, participants will review course materials (with the addition of the loneliness content for those assigned to the loneliness content condition) online and complete questionnaires assessing changes in various outcomes over time.

DETAILED DESCRIPTION:
Depression and anxiety are prevalent mental health conditions that are frequently under-treated. To improve timely and effective psychological treatment, Internet-delivered Cognitive Behaviour Therapy (ICBT) has been developed as a scalable treatment option. ICBT delivers evidence-based therapeutic content via structured online lessons over the course of several months, teaching the same skills as face-to-face cognitive behaviour therapy. In routine practice, ICBT is typically accompanied by brief therapist guidance offered via secure messaging and/or phone calls.

In Saskatchewan, the Online Therapy Unit (OTU) offers ICBT as part of routine care for a range of mental health concerns. The flagship program is the Wellbeing Course, a transdiagnostic ICBT program targeting symptoms of depression and anxiety. Research shows this course is associated with substantial significant improvements in depression and anxiety that are maintained over time. Nevertheless, not all clients engage with or respond equally to treatment. Consequently, there is a need to explore enhancements to ICBT that may improve outcomes for clients receiving care in naturalistic settings.

Emerging research shows a strong association between depression, anxiety and loneliness. Consistent with these findings, OTU recently found that approximately 76% of past OTU clients who enrolled in the Wellbeing Course reported experiencing frequent loneliness. Notably, ICBT was found to reduce loneliness in addition to alleviating symptoms of depression and anxiety.

Previous studies have found that many OTU clients engage with supplementary resources provided alongside the Wellbeing Course to tailor the program to their individual needs. However, no research to date has examined whether individuals experiencing frequent loneliness derive added benefit from receiving targeted content addressing loneliness in the context of ICBT for depression and anxiety.

The present trial aims to address this gap by evaluating whether offering additional loneliness content alongside the Wellbeing Course leads to greater engagement, satisfaction and improved treatment outcomes among clients with frequent loneliness compared to those who complete the Wellbeing Course alone.

The study is a partially randomized controlled trial conducted within a naturalistic online ICBT clinic. Clients seeking treatment who met the eligibility criteria and reported elevated levels of loneliness (i.e., ≥ 6 on the UCLA loneliness scale) are considered for inclusion in the study. Due to practical constraints related to therapist workload and the volume of referrals, not all eligible clients will be enrolled. To manage this, a subset of eligible clients are randomly assigned to one of two study conditions: (1) the Wellbeing Course or (2) the Wellbeing Course plus a Loneliness Resource. Other eligible clients are assigned to receive the standard Wellbeing Course outside of the study protocol, depending on service capacity at the time of intake. These non-study clients are not included in the study analyses. This approach allowed for the evaluation of the loneliness resource while maintaining routine clinical operations and equitable service access. Therapist support will be offered alongside the Course to all eligible clients for 8 weeks, with the possibility of extended support (when requested and clinically indicated) up to 12 weeks. Moreover, a booster session will be offered 12 weeks after the start of treatment to help clients review their progress and explore techniques that can assist in addressing any difficulties they may encounter in maintaining their well-being. All clients who take part in the Wellbeing Course will be asked to complete primary outcome questionnaires at screening and weeks 4, 8, and 20. Primary outcomes will be loneliness, depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Saskatchewan resident,
* Aged 18 years or older,
* Self-reported difficulty with depression and/or anxiety,
* Access to a computer (or other appropriate device) and the Internet,
* Willingness to learn information and skills to self-manage mental health difficulties, and
* Total score on UCLA-3 is greater than 5 at screening

Exclusion Criteria:

* Current severe medical or psychiatric condition that requires immediate treatment (e.g. current mania or psychosis, actively suicidal or unable to keep themselves safe, medical condition requiring immediate surgery or other invasive treatment);
* Unable to read and understand English (All content is provided in English and staff is English speaking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale 3-item (UCLA-3) | Baseline (Screening), weeks 4, 8 and 20 from enrollment
  Measures loneliness. 3 items are measured on a 3-point Likert scale ranging from 1-3. Scores are summed into a total score ranging from 3 to 9, with higher scores indicating higher levels of perceived loneliness.
Patient Health Questionnaire - 9 (PHQ-9) | Baseline (Screening), weeks 1-8 and 20 from enrollment
  Tracking the change in depression symptoms. 9 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed with total scores ranging from 0 to 27. Higher scores are associated with higher depression severity.
Generalized Anxiety Disorder - 7 (GAD-7) | Baseline (Screening), weeks 1-8 and 20 from enrollment
  Tracking the change in anxiety symptoms. 7 items are measured on a 4-point Likert scale ranging from 0-3. Scores are summed into a total score ranging from 0 to 21, with higher scores indicating more severe self-reported levels of anxiety.

SECONDARY OUTCOMES:
Things You Do - 15 (TYD-15) | Baseline (Screening), weeks 4, 8, and 20 from enrollment
  A measure of behaviors associated with mental health. 15 items are measured on a 5-point Likert scale ranging from 0-4. Subscales include Routine, Thoughts, Social, Activity, and Goals. Scores are summed into subscale scores ranging from 0 to 12, and a total score ranging from 0 to 60, with higher scores indicating increased engagement in behaviours associated with mental health.
Lubben Social Network Scale - 6 items (LSNS-6) | Baseline (Screening), weeks 8 and 20 from enrollment
  A measure assessing perceived social network and support using 6 items, with two subscales (Family and Friendship). Each subscale contains 3-items, measured on a 6-point Likert scale ranging from 0-5. Items on each subscale are summed to produce a subscale score ranging from 0 to 15. A total scale score ranges from 0 to 30. Higher scores indicate greater perceived support in each subscale or global scale.
Brief Social Support Scale (BS-6) | Baseline (Screening) weeks 8 and 20 from enrollment
  The BS-6 is a measure of perceived social support, with two subscales (emotional-informational and tangible social support). Each subscale contains 3-items. The first three items of the scale assess perceived tangible support and the remaining three items assess perceived emotional-informational social support. Items are measured on a 4-point Likert scale ranging from 1-4, with subscale scores ranging from 3 to 12, and global scores ranging from 6 to 24. Higher scores indicate greater perceived social support.
Mini Social Phobia Inventory (Mini SPIN) | Baseline (Screening), weeks 8 and 20 from enrollment
  Measures symptoms of social anxiety. 3 items are measured on a 5-point Likert scale ranging from 0 to 4. Scored are summed into a total score ranging from 0-12, with higher scores indicating greater symptoms of social anxiety.
Work and Social Adjustment Scale (WSAS) | Baseline (Screening), weeks 8 and 20 from enrollment
  The WSAS is a measure of functional impairment experienced in different interpersonal and intrapersonal domains due to mental health. Includes 5 items rated on a 9-point Likert scale ranging from 0-8. Scores are summed to produce a total score between 0-40. Higher scores indicate greater impairment in functioning.
Treatment Credibility and Expectancy Questionnaire (CEQ) | Baseline (Screening) and week 4
  Measures treatment credibility and expectancy using 6 items, with two subscales. First three items correspond to the credibility subscale and the following three items correspond to the expectancy subscale. Items are measured on 9-point Likert scale ranging from 1-9. Subscale scores range from 3 to 27. Higher scores in each subscale indicate greater treatment credibility or treatment expectancy respectively
Treatment Satisfaction Questionnaire | Week 8
  A 15-item questionnaire used to assess satisfaction with treatment and negative effects experienced by clients during treatment. The questionnaire uses a combination of Likert scale [5-point (0-4) and 6-point (0-5)], open-ended, and dichotomous yes/no response options to gauge participants' perceptions of the course. The questionnaire has been developed by the research team. A total score is not produced for this measure.
Loneliness Content Satisfaction | Week 8
  A bespoke 4-item measure administered to clients in the Wellbeing Course plus Loneliness Resource arm. The questionnaire uses a combination of dichotomous yes/no, Likert scale, and open-ended response option items to understand participants perceptions of the content. The questionnaire was developed by the research team and no total score is produced.

OTHER OUTCOMES:
Mental Health Service Use | Baseline (Screening), 20 weeks from enrollment
  An 11-item questionnaire assessing different parameters of mental health service usage, including providers and mental health services participants have accessed within the past three months, medication participants took for mental health concerns, employment status, and workplace accommodation/disabilities accessed. The questionnaire has been developed by the research team and does not have a score at this time. The questionnaire uses a combination of Likert scale, open-ended, and dichotomous yes/no response options to gauge participants' mental health service use.
Homework Reflection Questionnaire | Weeks 2 to 8
  A 5-item questionnaire assessing week-to-week experience in the course, with items inquiring about the lesson participants worked on; effort exerted towards skills; helpfulness of lessons; and client successes, challenges and experiences over the previous week. A combination of checklist, Likert scale [7-point (1-7)], and open-ended response options are used to gauge participants' participation. The questionnaire is used for clinicians to monitor treatment. No overall score is produced.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No